CLINICAL TRIAL: NCT07010848
Title: The Efficacy of Core Stability Training in Rehabilitation of Patients After Hip Fracture and in Patients After Stroke
Brief Title: the Efficacy of Core Stability Training in Rehabilitation
Acronym: Omino
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7406
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Hip Fractures
MeSH Terms: conditions — Stroke; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Patients with hip fractures or after stroke doing core stability training with standardised phyisiotherapy
  Interventions: Other: Core stability training
- Sperimental Group: Patients with hip fractures or after stroke doing core stability training with the utlization of "Omino" approach.
  Interventions: Other: Core stability training

INTERVENTIONS:
Other: Core stability training — Core stability Training consists in the activation of trunk.

SUMMARY:
The goal of the study is to verify the efficacy of core stability training in rehabilitation of patients after hip fracture and in patients after stroke.

The study will compare one group using traditional rehabilitation and another one with the addiction of an approach named "Omino", which is a kind of "health education" for the patient to the use of "Core Stability".

ELIGIBILITY:
Inclusion Criteria:

* age:18/90
* hip fracture
* stroke
* Consensus released

Exclusion Criteria:

* MMSE<24
* Dementia
* No Trunk control
* no deambulation
* clinical reasons
* consensus not released.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study selects geriatric patients tha need rehabilitation after hip fracture and after stroke.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ability in deambulation | 1 year
  the goal of the study is to verify the increase of ability in deambulation.

CONTACTS AND LOCATIONS:
Overall Officials: maria chiara patriarca, Principal Investigator — Fondazione Policlinico universitario Agostino Gemelli IRCSS